CLINICAL TRIAL: NCT03748615
Title: The Efficiency of Computer Guided Ridge Splitting Using Piezosurgery in Horizontally Deficient Posterior Mandible
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, walla farhat mohamed, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CairoUimplant master course
Record Dates: First submitted 2018-11-14; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Edentulous Patients; Atrophic Posterior Mandible With Insufficient Width

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computer Guided ridge splitting in posterior mandible (Experimental): fabrication of a computer aided surgical guide and performing ridge splitting in posterior mandible using piezosurgery
  Interventions: Device: Computer Guided ridge splitting in posterior mandible

INTERVENTIONS:
Device: Computer Guided ridge splitting in posterior mandible — The computer guided ridge splitting for patients with atrophic posterior mandible and with residual bone width at least 3 to 5mm of residual ridge.
  The selected patients will be informed of the nature of the research work and informed consent will be signed.
  Radiographic examination included preoperative digital panoramic radiograph with 1:1 magnification for each patient as a primary survey to obtain an approximation of the available bone height and detect the presence of remaining roots and localized pathosis.
  Computer surgical guides are fabricated for partially edentulous patients using teeth and tissue as support for the guide.
  The same surgeon performed all surgeries. All surgical procedures were performed under strict aseptic conditions, all patients received nerve block local anesthesia (Articaine 4% 1:100 000 epinephrine).
  A crestal incision is made using No. 15 blade extending over the posterior mandible using computer guided surgical stent.
  no flap elevation .

SUMMARY:
The use of implants has significantly increased prosthetic options for edentulous patient. However, implant placement in the Posterior mandibular region is often hampered significantly by insufficient atrophic width limitations

DETAILED DESCRIPTION:
Ridge splitting technique causes lateral ridge expansion which creates new implant bed by longitudinal osteotomy, positioning buccal cortex laterally. The buccal cortex is positioned laterally to create space between buccal and lingual cortical plates, which is filled by an endosseous implant with or without any graft material limitations.

Ridge split technique is a very predictable procedure that can achieve substantial gains in horizontal ridge width of the edentulous posterior mandible without associated morbidity. This technique allows the clinician to augment the site and do the implant insertion in a single stage surgery, shortening the healing period drastically.

In the conventional ridge splitting technique, a complete flap is raised to allow adequate visibility of the bone defect which can result in disturbance of vascular supply and increase bone resorption rates. In this case report, a new innovative computer guided closed alveolar ridge splitting flapless technique has been advocated to avoid this disruption.

As Guided implant placement showed a statistically superior accuracy when they are compared with freehand placement after guided osteotomy Computer guided ridge splitting may have a superior accuracy than the freehand ridge splitting and may reduce the time of surgery, healing period and post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with edentulous posterior area of the mandible insufficient width less than 5m, Both sexes.
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems.
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.
* Immunodeficiency pathology, bruxism, stress situation (socially or professionally), emotional instability, and unrealistic aesthetic demands.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11-20 (Estimated); Primary Completion 2019-09-20 (Estimated); Study Completion 2019-11-20 (Estimated)

PRIMARY OUTCOMES:
Time of the procedure ,pain and edema | 4 month
  the time of the procedure will be measured numerical using visual analogue scan